CLINICAL TRIAL: NCT03023033
Title: Enhancing Retention in PMTCT/MNCH Services and Facility Delivery in Tabora, Tanzania
Brief Title: Supporting Attendance for Facility Delivery and Infant Health
Acronym: SAFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Glaser Pediatric AIDS Foundation (Other)
Collaborators: Population Council (Other); Ministry of Health, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EG0130
Record Dates: First submitted 2015-02-27; First posted 2017-01-18 (Estimated); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: HIV; AIDS
Keywords: PMTCT; MNCH
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clinic group 1 (Experimental): Clinics using SMS health promotion and reminder messages (mhealth messaging)
  Interventions: Behavioral: mHealth messaging
- Clinic group 2 (Experimental): Clinics using SMS health promotion and reminder messages + Clinics providing payment scaled to reflect typical transport costs to facility (transport payments)
  Interventions: Behavioral: Transport Payments
- Clinic group 3 (No Intervention): Services provided under the Ministry of Health standard care

INTERVENTIONS:
Behavioral: mHealth messaging — SMS appointment reminders and health messaging via mobile phones
  Arms: Clinic group 1
Behavioral: Transport Payments — A payment scaled to reflect the cost of typical return transport fare for residents of the clinic catchment area
  Arms: Clinic group 2

SUMMARY:
The goal of this proposed intervention study is to increase the proportion of HIV positive and HIV negative pregnant women who deliver in a facility, the proportion of HIV exposed infants (HEI) who receive nevirapine (NVP) within 48 hours of delivery, and the proportion of HEI who are bled for HIV polymerase chain reaction (PCR) deoxyribonucleic acid (DNA) testing within 8 weeks of age.

DETAILED DESCRIPTION:
Following a formative phase I, we propose in phase II to implement a three-group cluster-randomized study to test the effectiveness of short message service (SMS) reminders and notifications, [mobile health or mhealth] (group 1) and the combined effectiveness of SMS reminders/notifications and cash transfers (group 2) compared to the standard prevention of mother-to-child transmission (of HIV)/maternal, neonatal and child health, (PMTCT/MNCH) practices (group 3).

ELIGIBILITY:
Inclusion Criteria:

* Known or recently diagnosed HIV-positive in ANC or; Tested HIV-negative at ANC
* Plans to deliver in facility catchment area
* 18 years or older
* Able and willing to provide consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1505 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Attendance for Early infant diagnosis (EID) of HIV | 1 year
  Proportion of HIV-exposed infants (HEI) attending for early infant diagnosis of HIV (DBS collected) by 8 weeks
Early identification of HEI at Reproductive and Child Health (RCH) Clinic | 1 year
  Proportion of HEI identified early (48 hours,3 and 7 days) at RCH clinic
Antenatal care (ANC) visits | 1 year
  Proportion of pregnant women attending at least 4 ANC visits
Facility delivery | 1 year
  Proportion of pregnant women delivering in a health facility
Post natal care (PNC) visits | 1 year
  Proportion of post partum women attending PNC 48 hours, 3 and 7 days post delivery
Nevirapine (NVP) at delivery | 1 year
  Proportion of HEI given NVP at delivery

SECONDARY OUTCOMES:
Receipt of EID results | 1 year
  Proportion of HEI who received EID results by 12 weeks
HIV infected infants initiated on antiretroviral therapy (ART) | 1 year
  Proportion of HIV infected infants initiated on ART by 12 weeks of age
Time to EID | 1 year
  Time (days/weeks) from date of birth to attendance for EID
Time to receipt of EID results | 1 year
  Time (days/weeks) from date of birth to receipt of EID results
Time to treatment | ! year
  Time (days/weeks) from date of birth to initiation of ART

CONTACTS AND LOCATIONS:
Overall Officials: Godfrey Woelk, MCOMMH, PhD, Principal Investigator — Elizabeth Glaser Pediatric AIDS Foundation
Locations (1):
- Elizabeth Glaser Pediatric AIDS Foundation, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
The dataset has been given to the USAID, the study sponsor. There is a plan to made these data publically available from 2018
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The plan is for the data to become available in 2018
Access Criteria: Access criteria will be defined by USAID

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276